CLINICAL TRIAL: NCT07104734
Title: Evaluation of the Ergogenic Properties of Citrus Flavonoid Hesperetin: Investigating Exercise-induced Fatigue, Oxidative Stress, Inflammation, Muscle Damage Mechanisms, and Judo-specific Performance
Brief Title: Evaluation of the Ergogenic Properties of Hesperetin on Exercise-induced Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CMUH113-REC2-012
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Athletes
Keywords: Hesperetin; judo; exercise performance
MeSH Terms: interventions — hesperetin

STUDY DESIGN:
Intervention Model Description: This study recruited 20 healthy male and female participants aged 12 to 30 years with at least 5 years of judo training experience to participate in a single-blind, pre-post test trial. Participants will be randomly assigned to either the hesperetin (Hst) group or the placebo group. All participants must be free from chronic conditions such as heart disease and hypertension, and must not have experienced any serious lower limb musculoskeletal injuries within the past six months. Throughout the study period, participants will be required to maintain their regular daily routines and will be prohibited from consuming any other nutritional supplements or alcohol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Containing edible yellow No. 4, edible yellow No. 5, sucrose, silica, talc, oxidized starch, gelatin, magnesium stearate, and palm wax.
  Interventions: Other: Placebo (Placebo trial); Other: Hesperetin (Hesperetin trial)
- Hesperetin (Experimental): Each capsule containing 250 mg of Hesperetin
  Interventions: Other: Placebo (Placebo trial); Other: Hesperetin (Hesperetin trial)

INTERVENTIONS:
Other: Placebo (Placebo trial) — The Placebo capsule supplement was taken for 2 weeks (2 capsules per day)
Other: Hesperetin (Hesperetin trial) — The Hesperetin capsule supplement was taken for 2 weeks, with a daily dosage of 500 mg of Hesperetin (equivalent to 2 capsules per day, each containing 250 mg of Hesperetin and 50 mg Pycnogenol®).

SUMMARY:
Twenty young, healthy, physically active men and women (12~30 years) did a pre-post trial randomized into placebo or HST trials (500 mg/d for two weeks). HST supplementation enhanced endurance judo-specific performance and effectively attenuated exercise-induced fatigue, oxidative stress, inflammatory response, and muscle damage.

DETAILED DESCRIPTION:
Participants in this study will be assigned identification numbers and randomly allocated to either the hesperetin (Hst) trial or the placebo trial. Seven days before the formal exercise performance test, all participants will undergo a maximal oxygen uptake (VO₂max) test using a cycle ergometer. The judo simulation consists of four consecutive 4-minute matches, each separated by a 30-minute rest. Participants will supplement with either placebo or Hst (500 mg/day) for 2 weeks. They are required to fast for 12 hours before the test day. On the experimental day, participants consume a light meal (300 kcal) and intake of either the placebo or Hst capsule, then rest for 1 hour. Afterward, participants perform a 15-minute judo-specific warm-up. All participants are required to complete all three matches. To standardize the judo simulation, opponents will be matched so that weight differences do not exceed 10%. Between the 30-minute rest time, blood samples will be collected and judo-specific physical performance will be evaluated. Immediately following the recovery period of the fourth match, the Special Judo Fitness Test (SJFT) will be evaluated. Judo-specific physical performance assessments will include grip strength, Counter Movement Jump (CMJ), and 10-second Wingate test.

ELIGIBILITY:
Inclusion Criteria:

* Judo athletes aged 12 to 30 years with at least 5 years of judo training experience.

Exclusion Criteria:

* All participants must be free from chronic conditions such as heart disease and hypertension, and must not have experienced any serious lower limb musculoskeletal injuries within the past six months.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Special Judo Fitness Test (SJFT) | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  The Special Judo Fitness Test (SJFT) was developed by Sterkowicz (1995) and has been validated through multiple studies demonstrating its objectivity, reliability, and validity. The SJFT consists of a task in which the athlete must throw a partner as many times as possible using maximum effort. The test is divided into three intervals: 15 seconds, 30 seconds, and 30 seconds, with 10-second rest periods in between. During each interval, the subject is verbally encouraged to perform as many throws as possible using the ippon-seoi-nage technique, with the throwing partners positioned 6 meters apart. After the test, heart rate (HR) is recorded immediately and again one minute post-exercise. The SJFT index is calculated based on the total number of throws and heart rate data using the following formula: SJFT Index = (Final HR [bpm] + HR at 1 minute post-test [bpm] / Total Number of Throws.
Upper Body Grip Strength Test | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  Grip strength will be measured using a handgrip dynamometer (SHM-18) to assess upper limb muscle strength. First, the examiner instructs the participant to let both arms hang naturally by the sides of the body. The grip span of the dynamometer is then adjusted so that the second knuckle of the index finger forms a right angle when gripping the handle. Once the correct posture is confirmed, the test begins.Grip strength will be measured on both the dominant and non-dominant hands. After completing one side and recording the value, the device is reset to zero, and the participant rests for 30 seconds before testing the other hand. During the test, the dynamometer must not come into contact with the body.Each hand is tested twice, and the maximum value (measured in kilograms) from the two trials on each side is recorded as the reference score.
Lower Limb Explosive Power - Countermovement Jump (CMJ) | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  The CMJ is used to assess lower limb maximal strength, explosive power, and speed. The CMJ test will be conducted using a sports performance measurement system to evaluate participants' lower limb explosive power. Under the guidance of the tester, participants will stand upright with knees fully extended, feet approximately shoulder-width apart, and hands placed on their waist to restrict arm swing, isolating lower limb performance.Participants will perform two maximal-effort jumps, with a 1-minute rest between attempts. The best jump height will be recorded as the test result. During the test, upon the tester's "start" command, participants will perform a rapid downward (countermovement) action to a self-selected depth, immediately followed by a maximal vertical jump.
10-Second Anaerobic Power Test | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  The test will be conducted using a stationary Monark 894E cycle ergometer. During the recovery period after each simulated judo match, participants will begin pedaling at a cadence of 60 rpm. The tester will then count down "3, 2, 1," and upon the "Go" command, participants will pedal at maximal effort and speed for 10 seconds. After completing the 10-second sprint, participants will continue pedaling at 60 rpm for a cooldown period as instructed by the tester to prevent dizziness caused by sudden cessation of exercise.Each participant will complete one 10-second anaerobic power test during the recovery period of each judo match. Anaerobic power indicators include peak power (occurring within the first 3 to 5 seconds of the test), total power output (W), and relative power output normalized to body weight (W/kg). The resistance load for the Wingate anaerobic power test is set at body weight (kg) × 0.75.
Assessment of the profile of mood state (POMS) | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  POMS brief was chosen for this study to evaluate the mood of individuals. After the TTE, participants completed the form, and their responses were analyzed using simple statistics. The results were shown in six dimensions, one positive: (1) vigor; and five negatives: (2) tension, (3) depression, (4) anger, (5) fatigue and (6) confusion.
Clinical Biochemistry of muscle damage biomarkers | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  Blood samples were collected at five different time points (15 min before the beginning (S), after each match (Match 1~3), and immediately (E) after the Special Judo Fitness Test. The concentrations of muscle damage markers creatine kinase (CK), myoglobin, and high-sensitivity C-reactive protein (hs-CRP) were measured using commercial assay kits (San Diego, CA, USA) and enzyme-linked immunosorbent assay (ELISA) with a microplate reader (Tecan GENios, A-5082, Austria). Absorbance was measured at 450 nm, 505 nm, and 572 nm, respectively. The concentrations of CK, myoglobin, and hs-CRP in serum samples were determined based on standard curves.
Clinical Biochemistry of oxidative stress | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  Blood samples were collected at five different time points (15 min before the beginning (S), after each match (Match 1~3), and immediately (E) after the Special Judo Fitness Test. The oxidative stress markers, including total antioxidant capacity (TAC), malondialdehyde (MDA), and thiobarbituric acid reactive substances (TBARS), were measured using commercial assay kits (Sigma, St.) and enzyme-linked immunosorbent assay (ELISA) with a microplate reader (Tecan GENios, A-5082, Austria). Absorbance was measured at 532 nm and 570 nm, and the concentrations of TAC, MDA, and TBARS in serum samples were determined based on standard curves.
Clinical Biochemistry of metabolic markers and safety assessment | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  Blood samples were collected at five different time points (15 min before the beginning (S), after each match (Match 1~3), and immediately (E) after the Special Judo Fitness Test. The metabolic markers glucose, non-esterified fatty acid (NEFA), and triglycerides (TG) were analyzed using commercial assay kits (WAKO NEFA, Germany) and measured with a fully automated biochemical analyzer (7020, Hitachi Science Systems, Ltd., Ibaraki, Japan). For safety assessment, GOP and GPT levels were determined using enzymatic analysis with commercial assay kits (Sigma, St.) and enzyme-linked immunosorbent assay (ELISA) on a microplate reader (Tecan GENios, A-5082, Austria). Absorbance was measured at 595 nm, and the concentrations of GOP and GPT in serum samples were calculated based on standard curves.
Clinical Biochemistry of cytokines | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  Blood samples were collected at five different time points (15 min before the beginning (S), after each match (Match 1~3), and immediately (E) after the Special Judo Fitness Test. The cytokines interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-α) were measured using commercial assay kits (Bio-Legend Inc., No. 430207, San Diego, CA, USA) and enzyme-linked immunosorbent assay (ELISA) with a microplate reader (Tecan GENios, A-5082, Austria). Absorbance was read at wavelengths of 450 nm and 570 nm, and the concentrations of IL-6 and TNF-α in serum samples were determined based on standard curves.
Clinical Biochemistry of stress markers | Including for 2 days in both pre-post test trials (which lasts around 2 weeks).
  Blood samples were collected at five different time points (15 min before the beginning (S), after each match (Match 1~3), and immediately (E) after the Special Judo Fitness Test. The stress markers catecholamine, cortisol, and testosterone were analyzed using commercial assay kits (San Diego, CA, USA) and measured with an enzyme-linked immunosorbent assay (ELISA) reader (Tecan GENios, A-5082, Austria). Absorbance was measured at 450 nm, 505 nm, and 572 nm, respectively. The concentrations of catecholamine, cortisol, and testosterone in serum samples were determined based on standard curves.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Piao Tsao, Study Chair — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No